CLINICAL TRIAL: NCT01018030
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Group, Multi-centre, 2-week Treatment Study to Evaluate the Safety and Efficacy of Fluticasone Furoate Nasal Spray 110 mcg in the Treatment in the Treatment of Uncomplicated Acute Rhinosinusitis in Adults and Adolescents >= 12 Years of Age
Brief Title: Dose Finding Study of Fluticasone Furoate Nasal Spray for Uncomplicated Acute Rhinosinusitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 113203
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Results first posted 2011-04-12 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Sinusitis, Acute
Keywords: uncomplicated acute rhinosinusitis; fluticasone furoate; sinusitis
MeSH Terms: conditions — Sinusitis | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- FFNS 110 mcg QD (Experimental)
  Interventions: Drug: FFNS 110 mcg QD
- FFNS 110 mcg BID (Experimental)
  Interventions: Drug: FFNS 110 mcg BID
- Placebo Nasal Spray (Placebo Comparator)
  Interventions: Drug: Placebo Nasal Spray

INTERVENTIONS:
Drug: FFNS 110 mcg QD — Active Nasal Spray (AM) and Placebo Nasal Spray (PM)
  Arms: FFNS 110 mcg QD
Drug: FFNS 110 mcg BID — Active Nasal Spray (AM) and Active Nasal Spray (PM)
  Arms: FFNS 110 mcg BID
Drug: Placebo Nasal Spray — Placebo Nasal Spray (AM) and Placebo Nasal Spray (PM)
  Arms: Placebo Nasal Spray

SUMMARY:
The purpose of this study is to assess the safety and efficacy of fluticasone furoate nasal spray (FFNS), without the use of an antibiotic, in the treatment of adult and adolescent subjects who are 12 years of age and older with uncomplicated acute rhinosinusitis (ARS).

DETAILED DESCRIPTION:
- Rationale - Acute rhinosinusitis (ARS) is a condition caused by inflammation of the nose and the paranasal sinuses that generally lasts up to 4 weeks. Despite ARS being a self-limiting condition, untreated or inadequately treated sinus infection can lead to the development of complications. Uncomplicated ARS is a subset of ARS and is distinguished from the common cold by the persistence or the worsening of sinus inflammation after the usual period for recovery of viral infection of the nasal cavity (i.e., 10 days). Clinically the difference is based on the following criteria: symptoms are present at least 10 days but less than 4 weeks beyond the onset of upper respiratory symptoms OR symptoms worsen after 5 days from their onset.

In the primary care settings, ARS is often treated empirically with antibiotics although they are shown to provide limited benefit in the uncomplicated ARS population. Alternatively, the use of an intranasal corticosteroid (INS) to control symptoms of uncomplicated ARS is plausible based on clinically proven ability to reduce inflammation and mucosal swelling.

This study is a phase II study.

* Objective - The objective of this study is to evaluate the safety and efficacy of two doses of FFNS (110 mcg once daily and 110 mcg twice daily) compared to placebo as monotherapy in the treatment of adult and adolescent subjects 12 years of age and older with uncomplicated ARS.
* Study Design - This is a randomized, double-blind, placebo controlled, parallel group, multi-centre, 2-week treatment study. The study includes a 2-week post-treatment follow-up period.

Approximately 720 subjects will be randomized to one of three treatment groups for a period of 14 days: FFNS 110 mcg QD, FFNS 110 mcg BID, and placebo nasal spray.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Outpatient
3. Age (>= 18 years at Visit 1 for Russia, Ukraine, and Germany; >= 12 years at Visit 2 for all other countries)
4. Diagnosis of uncomplicated acute rhinosinusitis
5. Ability and willingness to comply with study procedures and restrictions.
6. Male or eligible female - Female subjects should not be enrolled if they plan to become pregnant during the time of study participation; To be eligible for entry into the study, females of childbearing potential must commit to the consistent and correct use of an acceptable method of birth control.
7. Literate

Exclusion Criteria:

1. Based on the investigator's clinical judgement, subject has fulminant bacterial rhinosinusitis during the screening period including Visits 1 and 2.
2. A history of acute rhinosinusitis within 12 weeks prior to the current episode as determined by the investigator
3. Current or a history of other sinonasal conditions (e.g., chronic or recurrent rhinosinusitis, non-allergic rhinitis) within 3 years prior to Visit 1 as determined by the investigator
4. Symptomatic perennial or seasonal allergic rhinitis prior to ARS episode, or allergy to seasonal allergens likely to be present during the study period (as determined by documented skin prick test or in vitro blood test).
5. Significant concomitant medical conditions
6. Subjects with planned elective surgery, vacation or other event during the study period which could prevent the subject from participating in the study according to protocol specifications
7. Use of antibiotics within 30 days prior to Visit 1 for sinopulmonary infections.
8. Use of antiviral medications such as zanamivir and oseltamivir within 30 days prior to Visit 1
9. Use of analgesics or antipyretics within 1 day prior to Visit 1
10. Known hypersensitivity or allergy to corticosteroids or any excipients in the product
11. Use of corticosteroids, defined as:
12. Use of any other medications that may affect nasal symptoms
13. Use of immunosuppressive medications eight weeks prior to screening and during the study
14. Immunotherapy
15. Use of any medications that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4, including ritonavir and ketoconazole
16. Clinical trial/experimental medication experience
17. Positive pregnancy test or inconclusive pregnancy test or female who is breastfeeding
18. Affiliation with investigational site
19. Current tobacco use
20. Chicken pox or measles

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2010-01-06; Primary Completion 2010-07-01 (Actual); Study Completion 2010-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (75):
- Bulgaria (3):
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (20):
  - GSK Investigational Site, Chilliwack, British Columbia
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Ajax, Ontario
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Woodstock, Ontario
  - GSK Investigational Site, Granby, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saskatoon, Saskatchewan
- Czechia (5):
  - GSK Investigational Site, Benešov
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
- GSK Investigational Site, Tallinn, Estonia
- Germany (13):
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Ketzin, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Duisburg, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Delitzsch, Saxony
  - GSK Investigational Site, Schmölln, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Netherlands (6):
  - GSK Investigational Site, Almere Stad
  - GSK Investigational Site, Beek
  - GSK Investigational Site, Etten-Leur
  - GSK Investigational Site, Losser
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Woerden
- Norway (7):
  - GSK Investigational Site, Ålesund
  - GSK Investigational Site, Bekkestua
  - GSK Investigational Site, Elverum
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Hønefoss
  - GSK Investigational Site, Nesttun
  - GSK Investigational Site, Stavanger
- Poland (4):
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Zawadzkie
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- Spain (6):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Benidorm/Alicante
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Petrer/Alicante
  - GSK Investigational Site, Talavera de La Reina (Toledo)
- Sweden (4):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Lidingö
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Stockholm
- Ukraine (4):
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Symferopil
  - GSK Investigational Site, Zaporizhzhya

REFERENCES:
- [Background] Keith PK, Dymek A, Pfaar O, Fokkens W, Yun Kirby S, Wu W, Garris C, Topors N, Lee LA. Fluticasone furoate nasal spray reduces symptoms of uncomplicated acute rhinosinusitis: a randomised placebo-controlled study. Prim Care Respir J. 2012 Sep;21(3):267-75. doi: 10.4104/pcrj.2012.00039. PMID 22614920

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were randomized to a double-blind, placebo-controlled, parallel-group, 2-week treatment study to evaluate the safety and efficacy of fluticasone furoate nasal spray 110 micrograms (either once or twice daily) for the treatment of uncomplicated acute rhinosinusitis in adults and adolescent participants 12 years of age and older.
Groups:
- Placebo: Vehicle Placebo Nasal Spray administered twice daily (BD) for 14 days
- FFNS 110 mcg QD: Fluticasone Furoate Nasal Spray (FFNS) 110 micrograms (mcg) administered once daily (QD) in the morning and vehicle placebo nasal spray administered in the evening for 14 days
- FFNS 110 mcg BD: FFNS 110 mcg administered BD for 14 days
Period: Overall Study
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Started | 246 | 243 | 252
Completed | 227 | 232 | 239
Not Completed | 19 | 11 | 13
Not completed — Adverse Event | 10 | 5 | 5
Not completed — Withdrawal by Subject | 2 | 2 | 4
Not completed — Lost to Follow-up | 2 | 0 | 3
Not completed — Protocol Violation | 2 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Did Not Receive Study Drug | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD | Total
Number analyzed (Participants) | 245 | 240 | 252 | 737
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline Characteristics were collected in the Intent-to-Treat Population, comprised of all participants who were randomized and received at least one dose of double-blind study drug. One participant in the placebo group and three participants in the FFNS 110 mcg QD group did not receive any study treatment.
  Years | 39.1 (14.81) | 39.7 (15.64) | 39.0 (16.02) | 39.3 (15.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 143 | 148 | 169 | 460
  Male | 102 | 92 | 83 | 277
Race/Ethnicity, Customized [Number; unit: participants]
  White | 238 | 234 | 244 | 716
  Black | 3 | 0 | 3 | 6
  Other (Other than White and Black) | 4 | 6 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Daily Major Symptom Score (MSS) Over the Entire Treatment Period (Weeks 1-2)
Description: The MSS was calculated as the sum of 3 individual symptom scores for nasal congestion/stuffiness, sinus headache/pressure or facial pain/pressure, and postnasal drip. Daily MSS was calculated as the average of the morning (AM) and evening (PM) MSS. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe. The total score ranged from 0 to 9. Change from baseline was calculated as the daily MSS averaged over the entire treatment period minus daily MSS over the baseline period (defined as the average daily MSS over the last 3 days prior to randomization).
Time Frame: Baseline and entire treatment period (up to 2 weeks)
Population: Intent-to-Treat (ITT) Population: all randomized participants who received at least one dose of double-blind study drug. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 242 | 237 | 245
units on a scale | -2.97 (0.12) | -3.36 (0.13) | -3.33 (0.13)
Statistical Analysis 1: Comparison: Placebo vs FFNS 110 mcg QD; Test type: Superiority or Other; p = 0.008, ANCOVA; Least Squares Mean Difference = -0.386, 95% CI 2-sided [-0.67 to -0.10] — The estimation for least squares mean was adjusted for baseline value, country, allergic rhinitis status, age, and gender
Statistical Analysis 2: Comparison: Placebo vs FFNS 110 mcg BD; Test type: Superiority or Other; p = 0.014, ANCOVA; Least Squares Mean Difference = -0.357, 95% CI 2-sided [-0.64 to -0.07] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: First Time to Symptom Improvement
Description: Symptom improvement was defined as symptom scores less than or equal to 1 (i.e., mild or no symptoms) for all three major symptoms (nasal congestion/stuffiness, sinus headache/pressure or facial pain/pressure, and postnasal drip) on 2 consecutive 12-hour assessments. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe.
Time Frame: Entire treatment period (up to 2 weeks)
Population: ITT Population. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Median (Full Range); unit: days
Groups:
- Placebo: Vehicle Placebo Nasal Spray administered BD for 14 days
- FFNS 110 mcg QD: FFNS 110 mcg administered QD in the morning and vehicle placebo nasal spray administered in the evening for 14 days
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 243 | 239 | 247
days | 8 [1 to 14] | 7 [1 to 14] | 7 [1 to 14]

3. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in AM MSS
Description: Mean change from baseline in MSS for nasal congestion/stuffiness, sinus headache/pressure or facial pain/pressure, and postnasal drip as measured in the morning (AM) was calculated as the Week 1-2 value minus the baseline value. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe. The total score ranged from 0 to 9. Change from baseline in AM MSS was calculated as the AM MSS averaged over the entire treatment period minus the AM MSS over the baseline period (defined as the average AM MSS over the last 3 days prior to randomization).
Time Frame: Baseline and entire treatment period (up to 2 weeks)
Population: ITT Population. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 241 | 235 | 244
units on a scale | -3.1 (0.12) | -3.4 (0.12) | -3.3 (0.11)

4. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in PM MSS
Description: Mean change from baseline in MSS for nasal congestion/stuffiness, sinus headache/pressure or facial pain/pressure, and postnasal drip as measured in the evening (PM) was calculated as the Week 1-2 value minus the baseline value. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe. The total score ranged from 0 to 9. Change from baseline in PM MSS was calculated as the PM MSS averaged over the entire treatment period minus the PM MSS over the baseline period (defined as the average PM MSS over the last 3 days prior to randomization).
Time Frame: Baseline and entire treatment period (up to 2 weeks)
Population: ITT Population. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 242 | 236 | 242
units on a scale | -3.0 (0.12) | -3.4 (0.12) | -3.4 (0.12)

5. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in the Daily Nasal Congestion/Stuffiness Score
Description: Mean change from baseline was calculated as the Week 1-2 value minus the baseline value. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe. The score ranged from 0 to 3. Change from baseline in the daily nasal congestion/stuffiness score was calculated as the daily score averaged over the entire treatment period minus the daily score over the baseline period (defined as the average daily score over the last 3 days prior to randomization).
Time Frame: Baseline and entire treatment period (up to 2 weeks)
Population: ITT Population. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 242 | 237 | 245
units on a scale | -1.0 (0.04) | -1.1 (0.04) | -1.1 (0.04)

6. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in the AM Nasal Congestion/Stuffiness Score
Description: Mean change from baseline was calculated as the Week 1-2 value minus the baseline value. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe. The score ranged from 0 to 3. Change from baseline in the AM nasal congestion/stuffiness score was calculated as the AM score averaged over the entire treatment period minus the AM score over the baseline period (defined as the average AM score over the last 3 days prior to randomization).
Time Frame: Baseline and entire treatment period (up to 2 weeks)
Population: ITT Population. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 241 | 235 | 244
units on a scale | -1.0 (0.04) | -1.1 (0.04) | -1.1 (0.04)

7. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in the PM Nasal Congestion/Stuffiness Score
Description: Mean change from baseline was calculated as the Week 1-2 value minus the baseline value. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe. The score ranged from 0 to 3. Change from baseline in the PM nasal congestion/stuffiness score was calculated as the PM score averaged over the entire treatment period minus the PM score over the baseline period (defined as the average PM score over the last 3 days prior to randomization).
Time Frame: Baseline and entire treatment period (up to 2 weeks)
Population: ITT Population. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 242 | 237 | 242
units on a scale | -1.0 (0.04) | -1.1 (0.05) | -1.1 (0.04)

8. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in the Daily Sinus Headache/Pressure or Facial Pain/Pressure Score
Description: Mean change from baseline was calculated as the Week 1-2 value minus the baseline value. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe. The score ranged from 0 to 3. Change from baseline in the daily sinus headache/pressure or facial pain/pressure score was calculated as the daily score averaged over the entire treatment period minus the daily score over the baseline period (defined as the average daily score over the last 3 days prior to randomization).
Time Frame: Baseline and entire treatment period (up to 2 weeks)
Population: ITT Population. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 242 | 237 | 245
units on a scale | -1.1 (0.04) | -1.2 (0.05) | -1.2 (0.05)

9. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in the AM Sinus Headache/Pressure or Facial Pain/Pressure Score
Description: Mean change from baseline was calculated as the Week 1-2 value minus the baseline value. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe. The score ranged from 0 to 3. Change from baseline in the AM sinus headache/pressure or facial pain/pressure score was calculated as the AM score averaged over the entire treatment period minus the AM score over the baseline period (defined as the average AM score over the last 3 days prior to randomization).
Time Frame: Baseline and entire treatment period (up to 2 weeks)
Population: ITT Population. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 241 | 235 | 244
units on a scale | -1.2 (0.05) | -1.2 (0.05) | -1.2 (0.05)

10. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in the PM Sinus Headache/Pressure or Facial Pain/Pressure Score
Description: Mean change from baseline was calculated as the Week 1-2 value minus the baseline value. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe. The score ranged from 0 to 3. Change from baseline in the PM sinus headache/pressure or facial pain/pressure score was calculated as the PM score averaged over the entire treatment period minus the PM score over the baseline period (defined as the average PM score over the last 3 days prior to randomization).
Time Frame: Baseline and entire treatment period (up to 2 weeks)
Population: ITT Population. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 242 | 237 | 242
units on a scale | -1.1 (0.05) | -1.2 (0.05) | -1.2 (0.05)

11. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in the Daily Postnasal Drip Score
Description: Mean change from baseline was calculated as the Week 1-2 value minus the baseline value. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe. The score ranged from 0 to 3. Change from baseline in the daily postnasal drip score was calculated as the daily postnasal drip score averaged over the entire treatment period minus the daily postnasal drip score over the baseline period (defined as the average daily postnasal drip score over the last 3 days prior to randomization).
Time Frame: Baseline and entire treatment period (up to 2 weeks)
Population: ITT Population. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 242 | 237 | 245
units on a scale | -0.9 (0.05) | -1.0 (0.05) | -1.0 (0.04)

12. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in the AM Postnasal Drip Score
Description: Mean change from baseline was calculated as the Week 1-2 value minus the baseline value. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe. The score ranged from 0 to 3. Change from baseline in the AM postnasal drip score was calculated as the AM postnasal drip score averaged over the entire treatment period minus the AM postnasal drip score over the baseline period (defined as the average AM postnasal drip score over the last 3 days prior to randomization).
Time Frame: Baseline and entire treatment period (up to 2 weeks)
Population: ITT Population. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 241 | 235 | 244
units on a scale | -0.9 (0.05) | -1.1 (0.05) | -1.0 (0.04)

13. Secondary Outcome: Mean Change From Baseline Over the Entire Treatment Period in the PM Postnasal Drip Score
Description: Mean change from baseline was calculated as the Week 1-2 value minus the baseline value. Each individual symptom was scored on a scale of 0 to 3: 0=none; 1=mild; 2=moderate; 3=severe. The score ranged from 0 to 3. Change from baseline in the PM postnasal drip score was calculated as the PM postnasal drip score averaged over the entire treatment period minus the PM postnasal drip score over the baseline period (defined as the average PM postnasal drip score over the last 3 days prior to randomization).
Time Frame: Baseline and entire treatment period (up to 2 weeks)
Population: ITT Population. Participants with missing diary data at baseline or post-baseline were not included in this analysis.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 242 | 236 | 242
units on a scale | -0.9 (0.05) | -1.1 (0.05) | -1.0 (0.05)

14. Secondary Outcome: Number of Participants Who Require the Use of an Antibiotic Due to the Development of Fulminant Bacterial Rhinosinusitis (FBRS)
Description: Participants who required the use of an antibiotic due to the development of FBRS during the 2-week treatment period and the 2-week follow-up period were included in the analysis.
Time Frame: 4 weeks
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Number analyzed (Participants) | 245 | 240 | 252
participants | 7 | 7 | 7

ADVERSE EVENTS:
Arm/Group | Placebo | FFNS 110 mcg QD | FFNS 110 mcg BD
Serious Adverse Events (participants affected / at risk) | 0/245 | 0/240 | 1/252
Other Adverse Events (participants affected / at risk) | 41/245 | 41/240 | 46/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=245) | FFNS 110 mcg QD (N=240) | FFNS 110 mcg BD (N=252)
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=245) | FFNS 110 mcg QD (N=240) | FFNS 110 mcg BD (N=252)
Headache (Nervous system disorders) | 6 | 9 | 12
Sinusitis bacterial (Infections and infestations) | 6 | 6 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 3
Dizziness (Nervous system disorders) | 1 | 0 | 4
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 1 | 3
Bronchitis (Infections and infestations) | 2 | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 2
Nasal candidiasis (Infections and infestations) | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 1 | 1
Ear disorder (Ear and labyrinth disorders) | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 1
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal septum ulceration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 1 | 0
Oral pruritus (Gastrointestinal disorders) | 1 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Otosalpingitis (Ear and labyrinth disorders) | 0 | 1 | 0
Asthenia (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Glucose urine present (Investigations) | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.